CLINICAL TRIAL: NCT03739073
Title: Can we Predict COronary Resistance By EYE Examination ?
Brief Title: Can we Predict COronary Resistance By EYE Examination ? (COREYE)
Acronym: COREYE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_0301; 2018-A01181-54 (Other: ANSM)
Record Dates: First submitted 2018-11-05; First posted 2018-11-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with coronary arterial indication (Experimental): A fundus oculi and an OCTA (angiography by tomography in optical coherence) examination will be performed for patients with intermediate stenosis of the left anterior descending artery (LDA).
  Interventions: Other: OCTA (angiography by tomography in optical coherence)

INTERVENTIONS:
Other: OCTA (angiography by tomography in optical coherence) — The study concerns patients with intermediate stenosis of the left anterior descending artery (LDA). A fundus oculi and an OCTA (angiography by tomography in optical coherence) examination will be performed; it's a non-invasive imaging test. OCT uses light waves to take cross-section pictures of your retina and then ophthalmological examination data will correlate with coronary angiography.

SUMMARY:
Prospective interventional study, open, non-comparative and non-randomized. The research concerns physiological parameters of the coronary and ocular blood circulation.

At the coronary level, the curves of pressure and Doppler flow will be extracted from ComboMap® (Philips). The coronary microvascular resistances, basal and hyperemic, will be determined by the average ratio of the distal pressure and flow.

At the ocular level, a fundus oculi and an OCTA (angiography by tomography in optical coherence) examination will be performed. The measures of the FFR and the coronary microvascular resistance will be determined by a guidewire allowing measures of pressure and by a guidewire allowing measures of Doppler flow (ComboWire®, Volcano), in 123 patients with intermediate stenosis of the left anterior descending artery (LDA). Topological parameters characterizing the retinal area and choriocapillaries will be determined by statistical approaches and mathematical morphology.

To establish a predictor of the coronary microvascular resistance from the eye vascular parameters, we shall use a non-linear regression by supervised machine learning. The main cardiovascular risk factors (hypertension, diabetes, dyslipidemia, age, sex) will be part of predetermined input features for the machine learning.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patient's ≥18 years of age with coronary arterial indication as usual and with proximal and / or mean IVA stenosis ≥ 50%.
2. Signed informed consent
3. Affiliation to the social security system

Exclusion Criteria:

1. Unstable Coronary Artery Disease
2. Atrial fibrillation
3. History of myocardial infarction <6 months in the territory of the proximal and / or mean IVA.
4. Asthma
5. Aortocoronary bypass surgery.
6. Collateral development at the level of the proximal and / or mean IVA.
7. Allergy to iodine, severe renal insufficiency.
8. Ametropia> = 6 diopters.
9. History of retinal ocular pathologies other than uncomplicated diabetic retinopathy and hypertensive retinopathy.
10. History of ophthalmic treatments such as macular or panretinal laser photocoagulation, intravitreal injection of anti-VEGF or cortisone.
11. Chronic glaucoma
12. Patients under guardianship or curators.
13. Pregnant or lactating women.
14. Patient's not affiliated to the French social security.
15. Persons placed under the protection of justice,
16. Subject participating in another research including an exclusion period still in progress at pre-inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Coronary microvascular resistance results (Combowire) | Day 1
  Estimed by Combowire During coronary angiography, coronary resistance will be measured by pressure and Doppler guides in patients with intermediate coronary stenosis according to the usual procedure.
  Correlation between results of Combowire® coronary microvascular resistance and OCTA ophthalmologic findings. A machine learning technique will be used to analyze this series of ocular data and to determine a predictor of post-treatment coronary microvascular resistance.
Coronary microvascular resistance results (OCTA) | Day 1
  Estimated by ophthalmological examinations data from OCTA. An examination of fundus of the eye will then be performed by optical coherence tomography angiography without injection PLEX Elite 9000.
  Correlation between results of Combowire® coronary microvascular resistance and OCTA ophthalmologic findings. A machine learning technique will be used to analyze this series of ocular data and to determine a predictor of post-treatment coronary microvascular resistance.

SECONDARY OUTCOMES:
angiographical stenosis | Day 1
  measurement will be determined by guide allowing measurements of pressure and spectral Doppler (Combowire®)
Fractional Flow Reserve (FFR) | Day 1
  measurement of FFR will be determined by guide allowing measurements of pressure and spectral Doppler (Combowire®)
coronary microvascular resistance (CFR) | Day 1
  measurement of CFR will be determined by guide allowing measurements of pressure and spectral Doppler (Combowire®)
microvascular resistance values | Year 1
  Microvascular resistances will be measured using (Combowire®). The values of these resistances will be compared between the patient groups according to their cardiovascular risk factor
total area of flow signal void on the choriocapillaris layer | Year 1
  The total area of flow signal void on the choriocapillaris layer will be calculated with help of MATLAB software and will be correlated with cardiovascular risk-factors

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hopital de la Croix Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Harbaoui, B. (2021). Arterial stiffness, physiology, and relevance of interventional cardiology procedures (Habilitation à diriger des recherches thesis). Université Claude Bernard Lyon 1. (Manuscript hosted by CREATIS/INSA Lyon; defense notice by Lyon 1).